CLINICAL TRIAL: NCT04876534
Title: Multicenter, Randomized, Observer-blind, Controlled Study of the Anti-IL-6 Receptor Antibody Tocilizumab (TCZ) or Methylprednisolone (MP) Treatment in Patients With Active Moderate-severe Graves' Orbitopathy
Brief Title: Tocilizumab in Active Moderate-severe Graves' Orbitopathy
Acronym: TOGO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Mauriziano Umberto I Hospital (Other); Istituto Auxologico Italiano (Other); Azienda Ospedaliera "Sant'Andrea" (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML39921
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves' orbitopathy; Graves' disease; Tocilizumab; Hyperthyroidism; Thyroid's disease
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Hyperthyroidism | interventions — tocilizumab; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Intervention Model Description: 32 patients with active moderate-severe GO treated with i.v. tocilizumab; 32 patients with active moderate-severe GO treated with i.v. methylprednisolone.
Who Masked: Care Provider
Masking Description: The ophthalmologist assessing the ophthalmic changes is blinded to the patient's treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (Experimental): 32 patients with active moderate-severe GO treated with i.v. tocilizumab; Tocilizumab weight adjusted, 8 mg/kg, 1 intravenous infusion every four weeks (+/- 72 hours) for 12 weeks
  Interventions: Drug: Tocilizumab 20 Mg/mL Intravenous Solution
- Methylprednisolone (Active Comparator): 32 patients with active moderate-severe GO treated with i.v. methylprednisolone; Methylprednisolone, 500 mg infusion weekly (+/- 48 hours) for 6 weeks, followed by 250 mg infusion weekly (+/- 48 hours) for another 6 weeks
  Interventions: Drug: MethylPREDNISolone Injectable Solution

INTERVENTIONS:
Drug: Tocilizumab 20 Mg/mL Intravenous Solution — Intravenous administration
  Other Names: Actemra
  Arms: Tocilizumab
Drug: MethylPREDNISolone Injectable Solution — Intravenous administration
  Other Names: Solumedrol
  Arms: Methylprednisolone

SUMMARY:
To treat patientis with active moderate-severe GO with the anti-IL6 receptor monoclonal antibody tocilizubam with the purpose of assesing the efficacy of therapy on active GO and on the proportion of patiens with inactivation and reactivation of disease (Primary Objective) Effect of therapy on disease progression, improvement of QoL, the degree of residual disease after the inflammatory phase and safety of treatment (Secondary Objective)

DETAILED DESCRIPTION:
1 Primary Endpoint:

1. Proportion of patients with CAS reduction of 3 points or disease inactivation (CAS<4) at 12 and 24 weeks

1.2 Secondary Endpoints:

1. Proportion of patients improved at 24 weeks as assessed by the EUGOGO composite ophthalmic score (see below paragraph#5)
2. Improvement of quality of life according to the GO-QoL questionnaire at 12 and 24 weeks.
3. Safety of tocilizumab therapy in patients with GO compared to Methylprednisolone, evaluated on the basis of the following endpoints: Incidence and severity of adverse events, with severity determined according to NCI CTCAE v5.0,
4. Changes of serum TSH receptor binding and stimulating antibodies, anti-TPO antibodies and serum concentrations of IL-6 and sIL-6 receptor at 12, 24 and 36 and 48weeks of follow up.
5. Proportion of patients with disease reactivation (CAS > or =4) during follow-up at 24-48 weeks.
6. Quantification of signs of residual motility abnormalities by motility tests and orbital imaging
7. Number of rehabilitative surgical interventions at the end of follow-up

2.Study Design and Methods

Randomized, single blind (ophthalmologist), controlled study, IIb phase. The study will be conducted in 5 National centres dedicated to the management of Graves' orbitopathy

The present study will randomize GO patients, euthyroid for at least 6-8 weeks, to two treatments:

1. Tocilizumab weight adjusted, 8 mg/kg, 1 intravenous infusion every four weeks (+/- 72 hours) for 12 weeks
2. Methylprednisolone, 500 mg infusion weekly (+/- 48 hours) for 6 weeks, followed by 250 mg infusion weekly (+/- 48 hours) for another 6 weeks

The enrollment period is approximately 24 months

3.Phases of the study

* Screening phase (-4/-2 to 0 weeks): involves 1 to 2 visits
* Treatment phase (0 to 12 weeks): assessments at baseline and every 4 weeks
* Observation phase (12 to 24 weeks): assessments every 6 weeks
* Follow up (24 to 48 weeks): assessments every 12 weeks

Data from week 24 are used to determine primary and secondary endpoints

4.Definition of improvement, worsening or no change of the secondary end point criteria*

1. Improvement, when at least two of the following outcome measures improve in one eye, without deterioration in any of the measure in either eyes: a) reduction in palpebral aperture by at least 3 mm; b) reduction in any of the class 2 signs of NOSPECS by at least 2 grades; c) reduction of proptosis by at least 2 mm; d) improvement of ≥8 degrees in any duction or in diplopia (Gorman score); e) improvement in CAS by at least 2 points
2. Worsening, when optic neuropathy or two of the following occur: a) increase in palpebral aperture by at least 3 mm; b) increase in any of the class 2 signs of NOSPECS by at least 2 grades; c) increase of proptosis by at least 2 mm; d) deterioration of ≥8 degrees in any duction or in diplopia (Gorman score); e) worsening in CAS.
3. No change, when there are no changes or changes smaller than the above defined parameters

5. Study population

5.1 Withdrawal Rules

1. Should patients become affected with any of the conditions outlined as exclusion criteria during the study period or follow-up, they will be withdrawn from the study
2. Should patients require administration of any of the medications listed in the exclusion criteria, according to prohibited medication rules, they will be withdrawn from the study.
3. Other reasons for study withdrawal are:

   1. refusal of continuing the study medication after having commenced it.
   2. diagnosis of major cardiovascular diseases or neoplasia once treatment has started.
4. If patients present with a severe complication of GO, i.e. progression to dysthyroid optic neuropathy due to unresponsiveness to treatment, they will be considertreatment failure and will undergo urgent surgical orbital decompression.

Patients have the right to voluntarily withdraw from the study at any time for any reason. In addition, the investigator has the right to withdraw a patient from the study at any time. Reasons for withdrawal from the study may include, but are not limited to, the following:

Patient withdrawal of consent

Study termination or site closure

Patient non-compliance, defined as failure to comply with protocol requirements as determined by the investigator or Sponsor

Every effort should be made to obtain information on patients who withdraw from the study. The primary reason for withdrawal from the study should be documented on the appropriate eCRF. If a patient requests to be withdrawn from the study, this request must be documented in the source documents and signed by the investigator. Patients who withdraw from the study will not be replaced.

5.2 Study Arms

Arm 1: 32 patients with active moderate-severe GO treated with i.v. tocilizumab

Arm 2: 32 patients with active moderate-severe GO treated with i.v. methylprednisolone.

5.3 Study Medications and Dosing Regimen

Tocilizumab, the IMP-test, will be supplied and distribute by Roche packed and labelled.

Upon delivery to the site, site personnel should check for damage and verify proper identity, quantity, integrity of seals and temperature conditions. Site personnel should report any deviations or product complaints to the study monitor upon discovery.

For information on the formulation and handling of tocilizumab see the SmPC and Investigator's Brochure

Methylprednisolone is the IMP-comparator,

For information on the formulation, packaging, and handling of MP, see the SmPC.

Arm 1. Tocilizumab: i.v. infusion of, weight adjusted, 8 mg/kg of TCZ every four weeks (+/- 72 hours) for 12 weeks.

Arm 2. Methylprednisolone (MP): i.v. infusion of 500 mg of MP weekly (+/- 48 hours) for 6 weeks, followed by i.v. infusion of 250 mg of MP one a week (+/- 48 hours) for 6 weeks

5.4 Study duration

Duration of the study: 3 years (2 years for enrollment and one year for follow up)

5.5 Study Discontinuation

The Sponsor has the right to terminate this study at any time. Reasons for terminating the study may include, but are not limited to, the following:

The incidence or severity of adverse events in this or other studies indicates a potential health hazard to patients

Patient enrollment is unsatisfactory

The Sponsor will notify the investigator if the Sponsor decides to discontinue the study.

5.6 Site Discontinuation

The Sponsor has the right to close a site at any time. Reasons for closing a site may include, but are not limited to, the following:

Excessively slow recruitment

Poor protocol adherence

Inaccurate or incomplete data recording

Non-compliance with the International Council for Harmonisation (ICH) guideline for Good Clinical Practice

No study activity (i.e., all patients have completed the study and all obligations have been fulfilled)

6. Statistical considerations and sample size calculation A sample size of 64 patients is planned to provide at least an 80% power if 32 patients per treatment arm were included for an anticipated (improvement) responder rate of 68% in steroid and 95% in tocilizumab treated patients, with a two-tail significance of 0.05.

No patients stratification is planned The calculation is based on the available literature on the significant decrease of the after rituximab and steroid therapy and after tocilizumab and placebo.

64 patients with active GO will be enrolled and an interim analysis of results will be carried out after the first 32 patients (16 in arm 1 and 16 in arm 2) will reach the 24 week endpoint.

All enrolled patients receiving at least one dose of study medication and withdrawing from the study for any reason will be analyzed as non-responder in an ITT population for the 24 weeks primary endpoint.

Statistical Analysis: repeated measures ANOVA and Spearman or Pearson rank test for clinical activity and severity scores; Wilcoxon rank sum test to assess differences between treatment groups; chi-square for response and relapse rates.

An interim analysis of results will be carried out after the first 16 enrolled patients in both arms reach 24 week point), in order to eventually plan for another study perhaps employing s.c. TCZ .

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female, 18-75 years old
3. Women of childbearing potential should use effective contraception (abstinence or use contraceptive methods with a failure rate of <1%) throughout study and for a minimum of 6 months after study drug therapy and must have a negative serum pregnancy test at screening
4. GO at first diagnosis or at the time of relapse of no more than 9 months' duration.
5. Patients with moderate-severe active GO (clinical activity score 4/10 assessed at the end of the screening period) untreated or previously treated with i.v. steroids withdrawn for at least 3 months.
6. Euthyroid for at least 6-8 weeks (serum free hormone concentrations within 20% of normal range), on either anti-thyroid medications (tyonamides) to control hyperthyroidism or L-thyroxine for replacement therapy for hypothyroidism.
7. Patients will also be allowed to stay on propranolol treatment for the control of tachycardia.

Exclusion Criteria:

1. Patients with sight-threatening Graves' orbitopathy (severe keratopathy, compression optic neuropathy and inflammatory optic neuropathy).
2. Treatment with any biological therapy at any time.
3. Previous oral or intravenous corticosteroid treatment in the last three months except for oral steroid not exceeding a cumulative dose of 1 gr.
4. Plasmapheresis within 90 days prior to Day 0.
5. Treatment with intravenous immunoglobulin.
6. Azathioprine more than 100 mg/day within 30 days before screening.
7. Administration of live vaccines given within 30 days prior to administration of (Day 0) or concurrently with tocilizumab (during study).
8. Splenectomy.
9. Subjects at risk of bleeding that threatens a vital organ.
10. History of a major organ transplant or hematopoietic stem cell/marrow transplant.
11. History of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
12. Required management of infections, as follows: currently on any suppressive therapy for a chronic infection, hospitalization for treatment of infection within 60 days before Day 0, use of parenteral antibiotics within 60 days before Day 0, use of oral antibiotics within 30 days before Day 0.
13. Pregnancy.
14. Patients with reproductive potential not willing to use an effective method of contraception throughout study and for a minimum of 6 months after study drug therapy
15. Breast feeding.
16. Previous history of intestinal ulceration or diverticulitis or diverticular disease.
17. Known unstable coronary artery disease.
18. Significant cardiac arrhythmias.
19. Severe congestive heart failure.
20. Other serious chronic illness (including nervous system disease, pulmonary disease including obstructive pulmonary disease, renal disease).
21. Active infection.
22. History of recurrent clinically significant infection or recurrent bacterial infections.
23. History of sarcoidosis.
24. Primary or secondary immunodeficiency.
25. History of IgE-mediated or non-IgE-mediated hypersensitivity.
26. Positive PPD or quantiferon without documentation of treatment for TB infection.
27. Denied consent to HIV testing.
28. Previous orbital radiotherapy
29. HBsAg positive test.
30. HBcAb positive test, regardless of HBsAb status, will undergo HBV DNA which, if positive, will be excluded.
31. Hepatitis C antibody positive test at screening.
32. Positive test for Human Immunodeficiency Virus (HIV) antibody at screening or historically.
33. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) greater or equal to 1.5x upper limit of normal (ULN).
34. Alkaline phosphatase and bilirubin>1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is<35%).
35. Grade 3 / 4 IgG deficiency and IgA deficiency (IgA < 10mg/dL).
36. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy including a previous anaphylactic reaction to parenteral administration contrast agents, human or murine proteins or monoclonal antibodies.
37. Major depression.
38. Evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.
39. Current drug or alcohol abuse or dependence.
40. White blood cells < 3.0 x 109/L (3000/mm3)
41. Absolute neutrophil count (ANC) < 2.0 x 109/L (2000/ mm3)
42. Absolute lymphocyte count < 0.5 x 109/L (500/ mm3)
43. Platelet count <100 x 109/L
44. Serum creatinine > 1.4 mg/dl (124 µmol/L) in female patients and > 1.6 mg/dl (141 µmol/L) in male patients
45. Hemoglobin <85 g/L (8.5 g/dL; 5.3 mmol/L)
46. Demyelinating disorders
47. Treatment with Methotrexate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-12-18 (Estimated); Study Completion 2023-12-18 (Estimated)

PRIMARY OUTCOMES:
Desease inactivation | at 12 and 24 weeks
  Proportion of patients with CAS reduction of 3 points or disease inactivation (CAS<4) at 12 and 24 weeks

SECONDARY OUTCOMES:
Desease improvement | 24 weeks
  Proportion of patients improved at 24 weeks as assessed by the EUGOGO composite ophthalmic score
Improvement of quality of life | at 12 and 24 weeks
  Improvement of quality of life according to the GO-QoL questionnaire at 12 and 24 weeks. All Go-QoL questions were scored as 'severely limited' (one point), a 'little limited' (two points), or 'not limited at all'(three points). The questions were transformed from 0 to 100 by the following formula: total score= (raw score- 8)/16 x100. Higher is the final score, better is health.
Incident of adverse events in tocilizumab therapy | from 0 to 12 weeks
  Safety of tocilizumab therapy in patients with GO compared to Methylprednisolone, evaluated on the basis of the following endpoints: Incidence and severity of adverse events, with severity determined according to NCI CTCAE v5.0,
Immunological changes | at 12, 24 and 36 and 48weeks of follow up
  Changes of serum TSH receptor binding and stimulating antibodies, anti-TPO antibodies and serum concentrations of IL-6 and sIL-6 receptor at 12, 24 and 36 and 48weeks of follow up.
Desease relapse | at 24-48 weeks
  Proportion of patients with CAS reduction of 3 points from baseline CAS or disease inactivation (CAS<4) at 12 and 24 weeks.
  The Clinical activated score (CAS) is a parameter to assess eye impairment in patients with GO. The maximum CAS value is 10.
Residual desease | at 48 weeks
  Quantification of signs of residual motility abnormalities by motility tests and orbital imaging
Rehabilitative therapy | at 48 weeks
  Number of rehabilitative surgical interventions at the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mario MS Salvi, MD, Principal Investigator — Fondazione IRCCS "Cà Granda" Ospedale Maggiore Policlinico
Locations (4):
- Italy (4):
  - Istituto Auxologico Italiano, Milan, MI
  - Azienda Ospedaliero, Universitaria Pisana, Pisa, PI
  - Azienda Ospedaliera "Sant'Andrea", Roma, RM
  - Mauriziano Umberto I Hospital, Torino, TO

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartalena L, Baldeschi L, Boboridis K, Eckstein A, Kahaly GJ, Marcocci C, Perros P, Salvi M, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). The 2016 European Thyroid Association/European Group on Graves' Orbitopathy Guidelines for the Management of Graves' Orbitopathy. Eur Thyroid J. 2016 Mar;5(1):9-26. doi: 10.1159/000443828. Epub 2016 Mar 2. PMID 27099835
- [Background] Campi I, Vannucchi G, Salvi M. THERAPY OF ENDOCRINE DISEASE: Endocrine dilemma: management of Graves' orbitopathy. Eur J Endocrinol. 2016 Sep;175(3):R117-33. doi: 10.1530/EJE-15-1164. Epub 2016 Mar 31. PMID 27032693
- [Background] Salvi M, Campi I. Medical Treatment of Graves' Orbitopathy. Horm Metab Res. 2015 Sep;47(10):779-88. doi: 10.1055/s-0035-1554721. Epub 2015 Sep 11. PMID 26361263
- [Background] Campi I, Tosi D, Rossi S, Vannucchi G, Covelli D, Colombo F, Trombetta E, Porretti L, Vicentini L, Cantoni G, Curro N, Beck-Peccoz P, Bulfamante G, Salvi M. B Cell Activating Factor (BAFF) and BAFF Receptor Expression in Autoimmune and Nonautoimmune Thyroid Diseases. Thyroid. 2015 Sep;25(9):1043-9. doi: 10.1089/thy.2015.0029. Epub 2015 Aug 13. PMID 26214745
- [Background] Salvi M, Vannucchi G, Curro N, Campi I, Covelli D, Dazzi D, Simonetta S, Guastella C, Pignataro L, Avignone S, Beck-Peccoz P. Efficacy of B-cell targeted therapy with rituximab in patients with active moderate to severe Graves' orbitopathy: a randomized controlled study. J Clin Endocrinol Metab. 2015 Feb;100(2):422-31. doi: 10.1210/jc.2014-3014. Epub 2014 Dec 15. PMID 25494967
- [Background] Salvi M. Immunotherapy for Graves' ophthalmopathy. Curr Opin Endocrinol Diabetes Obes. 2014 Oct;21(5):409-14. doi: 10.1097/MED.0000000000000097. PMID 25105999
- [Background] Curro N, Covelli D, Vannucchi G, Campi I, Pirola G, Simonetta S, Dazzi D, Guastella C, Pignataro L, Beck-Peccoz P, Ratiglia R, Salvi M. Therapeutic outcomes of high-dose intravenous steroids in the treatment of dysthyroid optic neuropathy. Thyroid. 2014 May;24(5):897-905. doi: 10.1089/thy.2013.0445. Epub 2014 Mar 6. PMID 24417307
- [Background] Vannucchi G, Covelli D, Campi I, Origo D, Curro N, Cirello V, Dazzi D, Beck-Peccoz P, Salvi M. The therapeutic outcome to intravenous steroid therapy for active Graves' orbitopathy is influenced by the time of response but not polymorphisms of the glucocorticoid receptor. Eur J Endocrinol. 2013 Nov 22;170(1):55-61. doi: 10.1530/EJE-13-0611. Print 2014 Jan. PMID 24128430
- [Background] Salvi M, Vannucchi G, Beck-Peccoz P. Potential utility of rituximab for Graves' orbitopathy. J Clin Endocrinol Metab. 2013 Nov;98(11):4291-9. doi: 10.1210/jc.2013-1804. Epub 2013 Sep 5. PMID 24009135
- [Background] Vannucchi G, Covelli D, Curro N, Dazzi D, Maffini A, Campi I, Bonara P, Guastella C, Pignataro L, Ratiglia R, Beck-Peccoz P, Salvi M. Serum BAFF concentrations in patients with Graves' disease and orbitopathy before and after immunosuppressive therapy. J Clin Endocrinol Metab. 2012 May;97(5):E755-9. doi: 10.1210/jc.2011-2614. Epub 2012 Mar 7. PMID 22399512
- [Background] Salvi M, Vannucchi G, Curro N, Introna M, Rossi S, Bonara P, Covelli D, Dazzi D, Guastella C, Pignataro L, Ratiglia R, Golay J, Beck-Peccoz P. Small dose of rituximab for graves orbitopathy: new insights into the mechanism of action. Arch Ophthalmol. 2012 Jan;130(1):122-4. doi: 10.1001/archopthalmol.2011.1215. No abstract available. PMID 22232486
- [Background] Salvi M, Vannucchi G, Campi I, Curro N, Dazzi D, Simonetta S, Bonara P, Rossi S, Sina C, Guastella C, Ratiglia R, Beck-Peccoz P. Treatment of Graves' disease and associated ophthalmopathy with the anti-CD20 monoclonal antibody rituximab: an open study. Eur J Endocrinol. 2007 Jan;156(1):33-40. doi: 10.1530/eje.1.02325. PMID 17218723
- [Background] Vannucchi G, Campi I, Bonomi M, Covelli D, Dazzi D, Curro N, Simonetta S, Bonara P, Persani L, Guastella C, Wall J, Beck-Peccoz P, Salvi M. Rituximab treatment in patients with active Graves' orbitopathy: effects on proinflammatory and humoral immune reactions. Clin Exp Immunol. 2010 Sep;161(3):436-43. doi: 10.1111/j.1365-2249.2010.04191.x. PMID 20529087
- [Background] Salvi M, Vannucchi G, Campi I, Curro N, Simonetta S, Covelli D, Pignataro L, Guastella C, Rossi S, Bonara P, Dazzi D, Ratiglia R, Beck-Peccoz P. Rituximab treatment in a patient with severe thyroid-associated ophthalmopathy: effects on orbital lymphocytic infiltrates. Clin Immunol. 2009 May;131(2):360-5. doi: 10.1016/j.clim.2008.12.005. Epub 2009 Feb 4. PMID 19195932
- [Background] Yanaba K, Bouaziz JD, Matsushita T, Magro CM, St Clair EW, Tedder TF. B-lymphocyte contributions to human autoimmune disease. Immunol Rev. 2008 Jun;223:284-99. doi: 10.1111/j.1600-065X.2008.00646.x. PMID 18613843
- [Background] Rowland SL, Leahy KF, Halverson R, Torres RM, Pelanda R. BAFF receptor signaling aids the differentiation of immature B cells into transitional B cells following tonic BCR signaling. J Immunol. 2010 Oct 15;185(8):4570-81. doi: 10.4049/jimmunol.1001708. Epub 2010 Sep 22. PMID 20861359
- [Background] Moore PA, Belvedere O, Orr A, Pieri K, LaFleur DW, Feng P, Soppet D, Charters M, Gentz R, Parmelee D, Li Y, Galperina O, Giri J, Roschke V, Nardelli B, Carrell J, Sosnovtseva S, Greenfield W, Ruben SM, Olsen HS, Fikes J, Hilbert DM. BLyS: member of the tumor necrosis factor family and B lymphocyte stimulator. Science. 1999 Jul 9;285(5425):260-3. doi: 10.1126/science.285.5425.260. PMID 10398604
- [Background] Gilbert JA, Kalled SL, Moorhead J, Hess DM, Rennert P, Li Z, Khan MZ, Banga JP. Treatment of autoimmune hyperthyroidism in a murine model of Graves' disease with tumor necrosis factor-family ligand inhibitors suggests a key role for B cell activating factor in disease pathology. Endocrinology. 2006 Oct;147(10):4561-8. doi: 10.1210/en.2006-0507. Epub 2006 Jun 22. PMID 16794009
- [Background] Salvi M, Girasole G, Pedrazzoni M, Passeri M, Giuliani N, Minelli R, Braverman LE, Roti E. Increased serum concentrations of interleukin-6 (IL-6) and soluble IL-6 receptor in patients with Graves' disease. J Clin Endocrinol Metab. 1996 Aug;81(8):2976-9. doi: 10.1210/jcem.81.8.8768861.
- [Background] Campi I, Vannucchi GM, Minetti AM, Dazzi D, Avignone S, Covelli D, Curro N, Ratiglia R, Guastella C, Pignataro L, Beck-Peccoz P, Salvi M. A quantitative method for assessing the degree of axial proptosis in relation to orbital tissue involvement in Graves' orbitopathy. Ophthalmology. 2013 May;120(5):1092-8. doi: 10.1016/j.ophtha.2012.10.041. Epub 2013 Feb 8. PMID 23399378
- [Background] Perez-Moreiras JV, Gomez-Reino JJ, Maneiro JR, Perez-Pampin E, Romo Lopez A, Rodriguez Alvarez FM, Castillo Laguarta JM, Del Estad Cabello A, Gessa Sorroche M, Espana Gregori E, Sales-Sanz M; Tocilizumab in Graves Orbitopathy Study Group. Efficacy of Tocilizumab in Patients With Moderate-to-Severe Corticosteroid-Resistant Graves Orbitopathy: A Randomized Clinical Trial. Am J Ophthalmol. 2018 Nov;195:181-190. doi: 10.1016/j.ajo.2018.07.038. Epub 2018 Aug 4. PMID 30081019